CLINICAL TRIAL: NCT04901000
Title: Outcome of Local Versus General Anesthetic for Staged Carotid Endarterectomy Prior To CABG, Cohort Study
Brief Title: Outcome of LA Versus GA for Staged CEA Prior To CABG
Status: Completed | Type: Observational
Sponsor: Thomas Aherne (Other)
Collaborators: University Hospital Birmingham (Other)
Responsible Party: Sponsor-Investigator, Thomas Aherne, Site Investigator, National University of Ireland, Galway, Ireland
Organization: National University of Ireland, Galway, Ireland (Other)
Other Study IDs: University Hospital Birmingham
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Carotid Artery Diseases; Coronary Artery Disease; Stroke
MeSH Terms: conditions — Carotid Artery Diseases; Coronary Artery Disease; Stroke | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Carotid Endarterectomy under Local Anaesthetic Pre-CABG: Patients that underwent carotid endarterectomy under local anaesthetic prior to coronary artery bypass operations in staged fashion within 6 months.
  Interventions: Procedure: Carotid endarterectomy
- Carotid Endarterectomy under General Anaesthetic Pre-CABG: Patients that underwent carotid endarterectomy under general anaesthetic prior to coronary artery bypass operations in staged fashion within 6 months.
  Interventions: Procedure: Carotid endarterectomy

INTERVENTIONS:
Procedure: Carotid endarterectomy — Carotid endarterectomy prior to CABG operations either under Local Anaesthetic or under General Anaesthetic.

SUMMARY:
A retrospective analysis of all patients that underwent carotid endarterectomy (CEA) for stenotic disease - diagnosed at pre-operative investigation - prior to CABG as staged operation within 6- months.

The rate of postoperative stroke and complications was compared between CEA performed under Local anaesthetic (LA) to those performed under General anaesthetic (GA).

DETAILED DESCRIPTION:
The primary outcome was the rate of postoperative stroke in patients that had staged CEA prior to CABG. This was defined as CEA within a period of 4 weeks prior to CABG.

We retrospectively looked at those patients that fulfilled the inclusion criteria and had CEA performed either under LA (Group A) or under GA (Group B). We measured the 30 days' postoperative stroke rate as the main outcome. We also looked at the rate of intraoperative stroke.

Additionally, we assessed the rate for developing nerve injuries and/or hematoma postoperatively. Finally, we examined the risk for developing postoperative stroke in patients with bilateral significant carotid artery disease that underwent surgery in one side.

ELIGIBILITY:
Inclusion Criteria:

- All patients that had carotid endarterectomy performed in staged fashion within 6 months before a CABG operation.

Exclusion Criteria:

* Patients diagnosed with symptomatic carotid disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In-hospital patients referred by Cardiothoracic for carotid endarterectomy prior to CABG.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2011-10-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Stroke | 30 days
  a transient ischaemic attack (TIA), or a disabling stroke within 30 days of the carotid endarterectomy procedure.

SECONDARY OUTCOMES:
Major bleeding | 30 days
  Major haematoma was defined as a significant bleeding that required the patient to go back to theatre for a secondary procedure.
Minor bleeding | 30 days
  A minor hematoma was defined as bleeding that resulted in bruising and neck swelling without causing significant concerns to require a secondary procedur
Nerve injuries | 30 days
  Either neuropraxia that resolved with time or permanent injuries that resulted in disability.

IPD SHARING:
Plan to Share IPD: Undecided
Hospital records not to be shared, but raw data used for statistical analysis will be shared after removing identifiers.